CLINICAL TRIAL: NCT02826057
Title: The Complement Lectin Pathway in Patients Resuscitated After Cardiac Arrest
Brief Title: The Complement Lectin Pathway After Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 12345
Record Dates: First submitted 2016-06-16; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-06

CONDITIONS: Out-of-Hospital Cardiac Arrest; Post Cardiac Arrest Syndrome
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Post-Cardiac Arrest Syndrome | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 24 hour of targeted temperature management (Active Comparator): Patients resuscitated after cardiac arrest and treated with 24 hours of targeted temperature management (33 degree Celsius)
  Interventions: Other: Targeted temperature management (33 degree Celsius)
- 48 hour of targeted temperature management (Experimental): Patients resuscitated after cardiac arrest and treated with 48 hours of targeted temperature management (33 degree Celsius)
  Interventions: Other: Targeted temperature management (33 degree Celsius)

INTERVENTIONS:
Other: Targeted temperature management (33 degree Celsius)

SUMMARY:
This study includes comatose survivors of out-of-hospital cardiac arrest treated with 24 hours or 48 hours of targeted temperature management.

The overall aim is to evaluate the importance of plasma complement protein concentrations in patients resuscitated after out-of-hospital cardiac arrest and treated with 24 hours or 48 hours of targeted temperature management.

The specific aim is to evaluate:

* the concentration of plasma lectin pathway proteins the first, second and third day after cardiac arrest
* the relation between concentration of plasma lectin pathway proteins and mortality
* if prolonged targeted temperature management influences the concentration of plasma lectin pathway proteins

This study is a sub-study to the trial entitled: "Time-differentiated targeted temperature management (TTH48) (ClinicalTrials.gov Identifier: NCT01689077)"

The following Complement Lectin Pathway proteins will be measured: Mannan-Binding-Lectin, M-ficolin, H-ficolin, CL-L1, MASP-1, MASP-2, MASP-3, MAp19 and MAp44.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-Hospital Cardiac Arrest of presumed cardiac cause
* Return of spontaneous circulation (ROSC)
* Glasgow Coma Score < 8
* Age > 18 years and < 80 years

Exclusion Criteria:

* > 60 minutes from the circulatory collapse to ROSC
* Time interval > 4 hours from cardiac arrest to initiation of targeted temperature management
* Terminal illness
* Coagulation disorder
* Unwitnessed asystolia
* Cerebral performance category 3-4 before the cardiac arrest
* Severe persistent cardiogenic shock
* Pregnancy
* Persistent cardiogenic shock (systolic bloodpressure < 80 despite inotropic treatment)
* New apoplexy or cerebral hemorrhage
* Lack of consent from the relatives
* Lack of consent from the general practitioner
* Lack of consent from the patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
MASP-2 concentration in plasma | 48 hours

SECONDARY OUTCOMES:
MASP-2 concentration in plasma | 24 hours, 48 hours and 72 hours
MASP-2 concentration in plasma | 24 hours, 48 hours, 72 hours
  MASP-2 concentration in plasma compared with 30-day mortality
MASP-2 concentration in plasma | 24 hours to 72 hours
MASP-1 concentration in plasma | 24 hours, 48 hours and 72 hours
MASP-1 concentration in plasma | 24 hours to 72 hours
MASP-1 concentration in plasma | 24 hours, 48 hours, 72 hours
  MASP-1 concentration in plasma compared with 30-day mortality
MASP-3 concentration in plasma | 24 hours, 48 hours and 72 hours
MASP-3 concentration in plasma | 24 hours to 72 hours
MASP-3 concentration in plasma | 24 hours, 48 hours, 72 hours
  MASP-3 concentration in plasma compared with 30-day mortality
Mannan-Binding-Lectin concentration in plasma | 24 hours, 48 hours and 72 hours
Mannan-Binding-Lectin concentration in plasma | 24 hours to 72 hours
Mannan-Binding-Lectin concentration in plasma | 24 hours, 48 hours, 72 hours
  Mannan-Binding-Lectin concentration in plasma compared to 30-day mortality
MAp44 concentration in plasma | 24 hours, 48 hours and 72 hours
Map44 concentration in plasma | 24 hours to 72 hours
MAp44 concentration in plasma | 24 hours, 48 hours, 72 hours
  MAp44 concentration in plasma compared with 30-day mortality
MAp19 concentration in plasma | 24 hours, 48 hours and 72 hours
MAp19 concentration in plasma | 24 hours to 72 hours
MAp19 concentration in plasma | 24 hours, 48 hours, 72 hours
  MAp19 concentration in plasma compared with 30-day mortality
H-ficolin concentration in plasma | 24 hours, 48 hours and 72 hours
H-ficolin concentration in plasma | 24 hours to 72 hours
H-ficolin concentration in plasma | 24 hours, 48 hours, 72 hours
  H-ficolin concentration in plasma compared with 30-day mortality
M-ficolin concentration in plasma | 24 hours, 48 hours and 72 hours
M-ficolin concentration in plasma | 24 hours to 72 hours
M-ficolin concentration in plasma | 24 hours, 48 hours, 72 hours
  M-ficolin concentration in plasma compared with 30-day mortality
CL-L1 concentration in plasma | 24 hours, 48 hours and 72 hours
CL-L1 concentration in plasma | 24 hours to 72 hours
CL-L1 concentration in plasma | 24 hours, 48 hours, 72 hours
  CL-L1 concentration in plasma compared with 30-day mortality

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Department of Biomedicine, Aarhus University, Aarhus
  - Department of Anesthesiology and Intensive Care, Aarhus University Hospital, Aarhus
  - Department of Clinical Biochemistry, Aarhus University Hospital, Aarhus